CLINICAL TRIAL: NCT01900925
Title: Does Prescriptive Treatment of the Hips Improve Outcomes in Patients With Low Back Pain? A Randomized Controlled Trial
Acronym: HiLoBaS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regis University (Other)
Responsible Party: Principal Investigator, Michael Bade, Professor, Regis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC1937
Record Dates: First submitted 2013-07-07; First posted 2013-07-17 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Low Back Pain
Keywords: Low back pain, non-specific low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low back treatment only (pragmatic) (Active Comparator): 1. advise to stay active,
  2. discourage bed rest,
  3. appropriate medication use,
  4. reassurance.
  5. Short term use of manipulation/medication,
  6. supervised exercise,
  7. cognitive behavioral therapy,
  8. multidisciplinary treatment,
  9. termination of use of modalities.
  Interventions: Procedure: Pragmatic low back pain treatment
- LBP treatment and Hip treatment (Experimental): Group two will receive the same pragmatically applied, guideline-oriented treatment that is recommended from group 1. In addition, group 2 will receive prescriptive hip exercises that include 1) Clam Abduction exercises in sidelying, 2) Hip extension in quadruped, 3) a unilateral bridge, and the manual therapy treatment techniques of; 1) anterior to posterior mobilization of the hip with distraction, 2) long axis distraction of the hip and 3) posterior-anterior mobilization of the hip in prone.26 (See Appendix A for photos of the techniques and descriptions)
  Interventions: Procedure: Prescriptive Hip Exercises and Manual Therapy techniques; Procedure: Pragmatic low back pain treatment

INTERVENTIONS:
Procedure: Prescriptive Hip Exercises and Manual Therapy techniques — 1) Clam Abduction exercises in sidelying, 2) Hip extension in quadruped, 3) a unilateral bridge,and; 1) anterior to posterior mobilization of the hip with distraction, 2) long axis distraction of the hip and 3) posterior-anterior mobilization of the hip in prone
  Arms: LBP treatment and Hip treatment
Procedure: Pragmatic low back pain treatment — 1. advise to stay active,
  2. discourage bed rest,
  3. appropriate medication use,
  4. reassurance.
  5. Short term use of manipulation/medication,
  6. supervised exercise,
  7. cognitive behavioral therapy,
  8. multidisciplinary treatment,
  9. termination of use of modalities.
  Other Names: Low back pain treatment

SUMMARY:
There will be two groups of patients with low back pain (by randomization). Both groups will receive a pragmatic treatment approach by physical therapists for low back pain. One group will also receive a prescriptive treatment approach for both hips. The investigators feel that the additional of a standardized exercise program and stretching for the hips will improve outcomes in patients with mechanical low back pain.

DETAILED DESCRIPTION:
It has been suggested that treatment of the hips should improve outcomes in patients with mechanical low back pain. This has yet to be studied in a randomized controlled fashion or in a conservative venue. For this study, there will be two groups of patients with low back pain (by randomization). For inclusion into the randomized clinical trial, patients will need to be 18 years of age or older with mechanically producible LBP. They will require a minimum Modified Oswestry Disability Index score of 20% and a baseline pain score of >2.0/10 on the numeric analog scale for pain, and a within session change (improvement during the visit) in pain and/or range of motion during the assessment phase of the clinical examination. This finding has been advocated as an effective mechanism to determine if a patient is a candidate for manual therapy. Exclusion criteria will include the presence of any red flags (i.e., tumor, metabolic diseases, rheumatoid arthritis, osteoporosis, prolonged history of steroid use, etc.), or signs consistent with nerve root compression (reproduction of low back or leg pain with straight leg raise at less than 45°, muscle weakness involving a major muscle group of the lower extremity, diminished lower extremity muscle stretch reflex, or diminished or absent sensation to pinprick in any lower extremity dermatome). Other exclusion criteria include prior surgery to the lumbar spine and current pregnancy. Both groups will receive a pragmatic treatment approach by physical therapists for low back pain. One group will also receive a prescriptive treatment approach for both hips. The investigators will track the outcomes of disability (Oswestry), Pain (Numeric pain rating scale), and recovery at baseline, 2 weeks, and discharge. Our aims are to determine if differences in groups exist, with our primary outcome measure of ODI. The investigators feel that the additional of a standardized exercise program and stretching for the hips will improve outcomes in patients with mechanical low back pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Mechanically producible LBP.
* Minimum Modified Oswestry Disability Index score of 20%
* Minimum baseline pain score of >2.0/10 on the numeric analog scale for pain

Exclusion Criteria:

* Presence of any red flags
* Signs consistent with nerve root compression
* Prior surgery to the lumbar spine
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Modified Oswestry Disability Index | Baseline, 2 weeks, End of Intervention (Discharge)
  The Modified Oswestry Disability Index (ODI) will be used to measure disability, will serve as the primary outcome measure for the study, and consists of 10 questions each scored from 0 to 5, with higher scores indicating greater disability. A 50% reduction in the ODI or greater from baseline has been considered a clinically important outcome.

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale | Baseline, 2 weeks, End of Intervention (Discharge)
  An 11-point NPRS will be used to measure pain intensity. The scale is anchored on the left with the phrase "No Pain" and on the right with the phrase "Worst Possible Pain". NPRSs have been shown to be reliable and valid.32 Patients rate their current level of pain and their worst and least amount of pain experienced during the last 24 hours.
Recovery | End of Intervention (Discharge)
  A recent study has summarized the assortment of definitions associated with recovery.30 Recovery definitions associated with pain have ranged from 1) an absence of pain, to a maximal level of pain (e.g., 2/10 on an 11 point scale). Recovery definitions affiliated with function have included; 1) no functional dysfunction to 2) maximal level of functional loss (e.g., 20%/100% on a disability index). None have defined recovery in terms of a patient's perspective of recovery such as the patient acceptable symptom state (PASS) score. The PASS is the state beyond which patients consider their state as acceptable and are unlikely to seek further treatment.31 Thus, therapeutic success can be defined at the individual level (i.e., for each patient) as an improvement greater than minimum clinically acceptable score, or as achieving a state acceptable at the end of the care.31 For our study, recovery is defined as a "yes" (patients consider their state as acceptable) on the PASS at discharge.
Change in Global Rating of Change Score | 2 weeks and End of Intervention (Discharge)
  The fifteen-point global rating scale described by Jaeschke et al.,33 will be used. The scale ranges from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). The global rating scale will be administered at 4 visits, 1 month, and 6 months.
Change in Patient Satisfaction | 2 weeks and End of Intervention (Discharge)
  An 11-point patient satisfaction measure will be used to capture the patient's overall satisfaction with their intervention. The scale is anchored on the left with the phrase "Completely Dissatisfied" and on the right with the phrase "Completely Satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bade, PhD, PT, Principal Investigator — Regis University
Locations (1):
- Regis University, Denver, Colorado, United States